CLINICAL TRIAL: NCT00970723
Title: Role of High Blood Pressure and Sleep Apnea in Type 2 Diabetic Macular Edema
Brief Title: High Blood Pressure and Sleep Apnea in Diabetic Macular Edema
Acronym: OMHADIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P071227-AOM 08077
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic retinopathy; Macula edema; Sleep apnea; High blood pressure
MeSH Terms: conditions — Diabetic Retinopathy; Sleep Apnea Syndromes; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intensive treatment (Experimental): with a systematic screening for sleep apnea and/or uncontrolled high blood pressure, and intensified intervention on both anomalies if detected
  Interventions: Behavioral: high blood pressure treatment; Behavioral: sleep apnea treatment; Behavioral: diabetic macular edema treatment
- conventional treatment (Active Comparator): in accordance with national guidelines
  Interventions: Behavioral: diabetic macular edema treatment

INTERVENTIONS:
Behavioral: high blood pressure treatment — over one 14 month period: strongly recommended hygiene-dietetic measurements, complete assessment with ambulatory measurement of the blood pressure in D0, 3 and 12 months, a therapeutic strategy according to the results, and control every 3 months
  Arms: intensive treatment
Behavioral: sleep apnea treatment — over one 14 month period: complete assessment with night polysomnography in D0, 3 and 12 months, a therapeutic strategy according to the results, and control every 3 months
  Arms: intensive treatment
Behavioral: diabetic macular edema treatment — over one 14 month period: control every 3 months, treatments by laser (focal or grid) are authorized until 9 months, treatments by injections are authorized until 6 months

SUMMARY:
Macular edema remains a major cause of vision impairment in diabetic patients. Its pathogenesis is multifactorial and incompletely understood. Systemic factors seam to play a role in this pathogenesis, including high blood pressure. The objective of the study is to evaluate the effect of an intensified intervention on blood pressure and sleep apnea with that of conventional treatment in patients with type 2 diabetes and diabetic macular edema.

DETAILED DESCRIPTION:
Patients with type 2 diabetes and macular edema involving the center of the macula in both eyes will be randomly assigned to receive conventional treatment in accordance with national guidelines or to receive intensive treatment, with a systematic screening for sleep apnea and /or uncontrolled high blood pressure, and intensified intervention on both anomalies if detected. The primary outcome will be the percentage of patients having a sustained 50% or more-decrease in retinal thickening at 1 year. Secondary outcomes will be the percentage of patients having a 2 ETDRS lines or more-increase in visual acuity at one year, number of ocular interventions in each group, prevalence of sleep apnea and uncontrolled high blood pressure in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Patient with type 2 diabetes, aged 18 years or more
* Bilateral diabetic macular edema involving the center of the macula with central retinal thickness 300 µm or more

Exclusion Criteria:

* Patient with type 1 diabetes
* Tractional macular edema
* Patient with renal insufficiency : clearance of creatinin < 30 ml/min according to COCROFT or MDRD, patient under dialysis
* Other causes for macular edema (uveitis, epiretinal membrane)
* Proliferative diabetic retinopathy requiring panretinal photocoagulation at inclusion
* Cataract surgery or panretinal photocoagulation during the 6 months before inclusion, laser photocoagulation at the posterior pole or intra ocular steroid injection during the 3 months before inclusion
* Any ocular condition precluding access to the posterior pole, or ocular pathologies not related to diabetes (age related macular degeneration venous occlusion…)
* Previous vitrectomy in the eyes
* Pregnant or breast-feeding female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the percentage of patients having a sustained 50% or more-decrease in retinal thickening at 1 year, assessed with OCT in the study eye. | M13

SECONDARY OUTCOMES:
Percentage of patients having a 2 ETDRS lines or more-increase in visual acuity at one year in the study eye | M13
Number of ocular interventions (laser photocoagulation, intra ocular injections) in each group at one year in the study eye | M6-9
Progression of diabetic retinopathy in each group at one year according to the International DR classification in the study eye | M13
Comparison of blood pressure in each group at one year | M13

CONTACTS AND LOCATIONS:
Overall Officials: Pascale MASSIN, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (5):
- France (5):
  - Service d'ophtalmologie, Hôpital de la Vision, La Timone, Marseille, Bouches du Rhone
  - Service d'Ophtalmologie, Hôtel Dieu, Nantes, Loire Atlantique
  - Service d'Ophtalmologie, Hôpital Avicenne, Bobigny, Île-de-France Region
  - Hôpital Lariboisière, service d'Ophtalmologie, Paris, Île-de-France Region
  - Service d'Ophtalmologie IV, Hôpital des XV-XX, Paris, Île-de-France Region

REFERENCES:
- [Background] Paques M, Massin P, Sahel JA, Gaudric A, Bergmann JF, Azancot S, Levy BI, Vicaut E. Circadian fluctuations of macular edema in patients with morning vision blurring: correlation with arterial pressure and effect of light deprivation. Invest Ophthalmol Vis Sci. 2005 Dec;46(12):4707-11. doi: 10.1167/iovs.05-0638. PMID 16303968